CLINICAL TRIAL: NCT01935674
Title: Rosuvastatin Versus Protease Inhibitor Switching for Hypercholesterolaemia in HIV-infected Adults
Brief Title: Treatment With Rosuvastatin Versus Switching PI (Protease Inhibitor) in Patients HIV With High Cholesterol Levels
Acronym: SOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, Project manager, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOS
Record Dates: First submitted 2013-03-19; First posted 2013-09-05 (Estimated); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: HIV; Hypercholesterolaemia
Keywords: Hypercholesterolaemia; HIV; Rosuvastatin; Protease inhibitor switching
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Switch ritonavir-boosted PI (Experimental): Switch their existing ritonavir-boosted PI to another potent ART drug with lesser effects on serum cholesterol selected by the investigator.
  Interventions: Drug: Switch ritonavir-boosted PI
- Continue ritonavir-boosted PI+Rosuvastatin (Experimental): Continue ritonavir-boosted PI-based ART and commence rosuvastatin 10 mg daily (5 mg daily in Asian participants).
  Interventions: Drug: Continue Ritonavir-boosted PI+Rosuvastatin

INTERVENTIONS:
Drug: Switch ritonavir-boosted PI — Switch their existing ritonavir-boosted PI to another potent ART drug with lesser effects on serum cholesterol selected by the investigator.
  Arms: Switch ritonavir-boosted PI
Drug: Continue Ritonavir-boosted PI+Rosuvastatin — Continue ritonavir-boosted PI-based ART and commence rosuvastatin 10 mg daily (5 mg daily in Asian participants).
  Arms: Continue ritonavir-boosted PI+Rosuvastatin

SUMMARY:
To compare the effect of rosuvastatin to protease inhibitor switching on fasting total cholesterol over 12 weeks.

DETAILED DESCRIPTION:
To compare the effects of rosuvastatin to protease inhibitor switching on:

* Total cholesterol through week 12
* Safety parameters (HIV viral load, clinical adverse events, serious adverse events, laboratory adverse events, modifications to antiretroviral therapy)
* Quality of life (SF-12)
* Fasting LDL cholesterol (estimated with Friedewald equation unless triglycerides >400mg/dL, in which case LDL-C would be measured directly), HDL cholesterol, total : HDL cholesterol ratio, LDL particles sizes, triglycerides
* Fasting glucose and insulin
* Framingham cardiovascular risk score
* D:A:D 5-year estimated risk calculator

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive status
* Adults (≥18 years of age)
* Stable and well-tolerated combination ART including a ritonavir-boosted protease inhibitor for the previous 6 months
* HIV RNA <50 copies/mL for at least the preceding 3 months
* Fasting total cholesterol ≥5.5 mmol/L (>213 mg/dL)
* Framingham risk score ≥8% at 10 years OR diabetes mellitus OR a family history of premature coronary artery disease in a first-degree relative
* Provision of written, informed consent

Exclusion criteria:

* Any statin in the previous 12 weeks
* Previous statin-induced myopathy or hepatitis
* History of coronary artery disease, stroke or any other indication for the use of statin therapy (hyperlipidaemia: genetic, secondary or idiopathic)
* Concurrent use of:

  1. oral corticosteroids use other than for replacement therapy (i.e. prednisolone 5-7.5 mg, hydrocortisone 20-30 mg, cortisone acetate 25-37.5 mg daily)
  2. other immunosuppressive or immunomodulating drugs
* Contraindication to rosuvastatin therapy:

  1. liver transaminases >5 times the upper normal limit
  2. creatinine clearance <30 mL/min
  3. known myopathy
  4. current fibrate therapy
  5. known resistance to one or more "backbone" ART drugs
* No potent switch ART drug available to replace the current ritonavir-boosted protease inhibitor
* Known intolerance to rosuvastatin or the proposed switch ART drug
* Women attempting or likely to become pregnant, or who are pregnant or breast-feeding
* A patient with a history or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study, or interfere with the patient's participation for the full duration of the study
* Unable to complete study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Martinez, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain

REFERENCES:
- See also: Rosuvastatin vs. protease inhibitor switching for hypercholesterolaemia: a randomized trial — https://pubmed.ncbi.nlm.nih.gov/26987376/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between June 2012 and April 2014 across nine clinical sites in Australia and Spain, including hospitals and private HIV clinics. Recruitment targeted HIV-1-infected adults with controlled viral load and elevated cardiovascular risk, not currently on lipid-lowering therapy.
Pre-assignment Details: After providing informed consent, participants underwent a screening period of up to 14 days to confirm eligibility. This included fasting blood tests, cardiovascular risk assessment (Framingham score), and confirmation of stable ART. Participants were excluded prior to randomization if they did not meet inclusion criteria (e.g., cholesterol <5.5 mmol/L, low cardiovascular risk, or contraindications to study drugs). No washout or run-in period was required.
Period: Overall Study
Arm/Group | Switch Ritonavir-boosted PI | Continue Ritonavir-boosted PI+Rosuvastatin
Started | 20 | 23
Completed | 20 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants (N=43) were included in the baseline analysis population. No participants were excluded post-randomization, and all contributed data to the primary endpoint analysis (intention-to-treat population).
Groups:
- PI/r Switch Group: Switch their existing ritonavir-boosted PI to another potent ART drug with lesser effects on serum cholesterol selected by the investigator.
  Switch ritonavir-boosted PI: Switch their existing ritonavir-boosted PI to another potent ART drug with lesser effects on serum cholesterol selected by the investigator.
- Rosuvastatin: Continue ritonavir-boosted PI-based ART and commence rosuvastatin 10 mg daily (5 mg daily in Asian participants).
  Continue Ritonavir-boosted PI+Rosuvastatin: Continue ritonavir-boosted PI-based ART and commence rosuvastatin 10 mg daily (5 mg daily in Asian participants).
- Total: Total of all reporting groups
Arm/Group | PI/r Switch Group | Rosuvastatin | Total
Number analyzed (Participants) | 20 | 23 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (8.2) | 53 (8.7) | 55 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 20 | 22 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 22 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Total cholesterol [Mean (Standard Deviation); unit: mmol/L] | 6.0 (0.9) | 6.3 (1.4) | 6.2 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Total Cholesterol at 12 Weeks.
Description: The outcome was defined as the percentage change in fasting total cholesterol from baseline (week 0) to week 12. Fasting blood samples were collected after a 12-hour fast, and total cholesterol was measured in mmol/L. The percentage change was calculated for each participant and compared between the rosuvastatin and PI/r switch groups using an intention-to-treat analysis.
Time Frame: 12 weeks from baseline (week 0 to week 12)
Measure: Mean (Standard Deviation); unit: Percentage Change (%)
Arm/Group | PI/r Switch Group | Rosuvastatin
Number analyzed (Participants) | 20 | 23
Percentage Change (%) | 8.7 (10.8) | 21.4 (19.2)
Statistical Analysis 1: Comparison: PI/r Switch Group vs Rosuvastatin; Comparison of percentage change in fasting total cholesterol from baseline to week 12 between rosuvastatin and PI/r switch groups. Wilcoxon rank-sum test used. Study powered to detect a 15% difference with 80% power and α = 0.05. All participants included in intention-to-treat analysis; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney) — P-value from Wilcoxon rank-sum test; significance threshold set at α = 0.05. No adjustment for multiple comparisons; Two-sided test; analysis based on intention-to-treat population; Mean Difference (Net) = 12.7, 95% CI 2-sided [2.9 to 22.5]

2. Secondary Outcome: Total Cholesterol Through Week 12
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Safety Parameters (HIV Viral Load, Clinical Adverse Events, Serious Adverse Events, Laboratory Adverse Events, Modifications to Antiretroviral Therapy)
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Quality of Life (SF-12)
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Fasting LDL Cholesterol (Estimated With Friedewald Equation Unless Triglycerides >400mg/dL, in Which Case LDL-C Would be Measured Directly), HDL Cholesterol, Total : HDL Cholesterol Ratio, LDL Particles Sizes, Triglycerides
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Fasting Glucose and Insulin.
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Framingham Cardiovascular Risk Score (10-year Risk Estimate)
Description: The Framingham Risk Score is a sex-specific algorithm used to estimate the 10-year risk of developing cardiovascular disease (CVD), including coronary heart disease, stroke, peripheral artery disease, and heart failure. It is based on factors such as age, sex, total cholesterol, HDL cholesterol, systolic blood pressure, treatment for hypertension, smoking status, and diabetes.
  Scale Title: Framingham 10-Year Cardiovascular Risk Score Minimum Value: 0% Maximum Value: 100% Interpretation: Higher scores indicate a worse outcome, meaning a higher estimated risk of developing cardiovascular disease within 10 years.
Time Frame: Screening and week 12
Reporting Status: Not Posted

8. Secondary Outcome: D:A:D 5-year Estimated Risk Calculator.
Time Frame: Screening and week 12.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events were graded according to the Division of AIDS (DAIDS) adverse event grading table [23], and assigned causality; participants were directly asked about gastrointestinal and musculoskeletal events. Between-group adverse event rates were compared using the χ² test.
Arm/Group | PI/r Switch Group | Rosuvastatin
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/23
Other Adverse Events (participants affected / at risk) | 14/20 | 14/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PI/r Switch Group (N=20) | Rosuvastatin (N=23)
Unstable angina requiring coronary artery stenting (Cardiac disorders) | 0 (0) | 1 (1) — Occurred in rosuvastatin group; not related to study drug.
Tibial fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PI/r Switch Group (N=20) | Rosuvastatin (N=23)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) — Mild; more frequent in PI/r switch group
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) — Mild; only reported in PI/r switch group
Fatigue (General disorders) | 2 (2) | 0 (0) — Mild; only in PI/r switch group
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Mild; only in PI/r switch group.
Other (Investigations) | 6 (6) | 0 (0) — Includes various mild symptoms not otherwise specified.
Unespecified non drug-related events (General disorders) | 4 (4) | 13 (13)

LIMITATIONS AND CAVEATS:
Small, short-duration study with a homogeneous population. Not powered for clinical outcomes. Results may not generalize broadly.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-10-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT01935674/Prot_SAP_000.pdf